CLINICAL TRIAL: NCT07350174
Title: A Multicenter, Open-label, Randomized, Active-controlled, Phase 2a Study to Evaluate the Pharmacokinetics and Safety of Alpibectir/Ethionamide in Combination With the Standard Regimen in Patients With Tuberculosis Meningitis.
Brief Title: Phase 2a Trial of Alpibectir Plus Ethionamide for Tuberculosis Meningitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioVersys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlpE-TBM
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis Meningitis
Keywords: Tuberculosis, AlpE, Ethionamide, CSF, pharmacokinetics
MeSH Terms: conditions — Tuberculosis, Meningeal; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: HRZE (Active Comparator)
  Interventions: Drug: HRZE
- Group 2: HRZE plus Alpe375 (Experimental)
  Interventions: Drug: HRZE plus Alpe375
- Group 3: HRZE plud AlpE500 (Experimental)
  Interventions: Drug: HRZE plus AlpE500
- Group 4: HRZE plus AlpE625 (Experimental)
  Interventions: Drug: HRZE plus AlpE625

INTERVENTIONS:
Drug: HRZE — Isoniazid (5 mg/kg/day); Rifampicin (10 mg/kg/day); Pyrazinamide (30 mg/kg/day); Ethambutol (20 mg/kg/day).
  Arms: Group 1: HRZE
Drug: HRZE plus Alpe375 — isoniazid (5 mg/kg/day); rifampicin (10 mg/kg/day); pyrazinamide (30 mg/kg/day); ethambutol (20 mg/kg/day), Alpe375 (alpibectir (30 mg/day), ethionamide (375 mg/day))
  Arms: Group 2: HRZE plus Alpe375
Drug: HRZE plus AlpE500 — isoniazid (5 mg/kg/day); rifampicin (10 mg/kg/day); pyrazinamide (30 mg/kg/day); ethambutol (20 mg/kg/day), Alpe375 (alpibectir (30 mg/day), ethionamide (500 mg/day))
  Arms: Group 3: HRZE plud AlpE500
Drug: HRZE plus AlpE625 — isoniazid (5 mg/kg/day); rifampicin (10 mg/kg/day); pyrazinamide (30 mg/kg/day); ethambutol (20 mg/kg/day), Alpe375 (alpibectir (30 mg/day), ethionamide (625 mg/day))
  Arms: Group 4: HRZE plus AlpE625

SUMMARY:
AlpE is a novel drug combination under development for the treatment of TB, with several positive attributes for TBM, including rapid bactericidal activity. The current trial aims to assess the plasma and CSF PK, as well as the safety and tolerability of alpibectir and three doses of Eto in patients with newly diagnosed TBM. Additionally, we will investigate the effect of AlpE on the PK and efficacy of DTG during the first month of antiretroviral treatment (ART) for Human Immunodeficiency Virus (HIV)-positive patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 15 years and < 65 years
2. Diagnosis of TBM defined as "definite" or "probable", using criteria proposed by the Tuberculosis Meningitis International Research Consortium.

   * Definite TBM is defined by at least one of the following criteria: acid-fast bacilli (AFB) seen in CSF microscopy, positive CSF M. tuberculosis culture, or positive CSF M. tuberculosis commercial nucleic acid amplification test in the setting of symptoms suggestive of meningitis.
   * Probable TBM is defined using a modified Marais score* Probable TBM: total score* ≥ 12 when neuroimaging is available, or ≥ 10 when neuroimaging is not available. At least 2 points should come from CSF or 2 points from cerebral imaging criteria.

   (*see Appendix 2: Modified Marais Score)
3. Informed consent signed by the patient. For patients with Glasgow Coma Scale (GCS) < 15, the consent of a next of kin/relative will be required, in accordance with applicable local laws and regulations. Deferred consent will be obtained from the participant when their level of consciousness improves, and they have capacity to provide consent. For adolescents below the age of civil majority (as defined in each country), the consent of at least one parent or legal guardian and the assent of the adolescent will be required.

Exclusion Criteria:

1. Having received >14 days of HRZE TB treatment.
2. In people with HIV infection: use of antiretroviral treatment (ART) other than efavirenz- or dolutegravir-based.
3. Glasgow Coma Scale < 10.
4. Body weight measured or estimated: < 40 kg or > 90 kg or BMI > 40 kg/m2.
5. Renal failure (eGFR < 30 mL/min, calculated by CKD-EPI formula).
6. Alanine aminotransferase (ALT) > 5 times the Upper Limit of Normal.
7. Clinical evidence of liver failure or decompensated cirrhosis.
8. For women of childbearing potential, one or more of the following:

   1. Being pregnant, breast-feeding, or intending to breast-feed or conceive a child during the study or within 30 days after the end of treatment visit (D56), OR;
   2. Not willing or able to use highly effective contraceptive methods (as defined per Appendix 7) starting at screening and continuing until 30 days after the end of treatment visit (D56).
9. For male participants: intending to conceive a child or not willing or able to consistently use a barrier method e.g. condoms during all sexual activity from inclusion until 90 days after the end of treatment visit (D56).

   Note: Male participants should be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse.
10. Documented Mtb resistance to rifampicin.
11. Positive Gram-stain, bacterial culture other than Mtb or cryptococcal antigen in the CSF.
12. For HIV positive patients: Presence of cryptococcal antigen in the blood.
13. Inability to collect CSF or contraindication to lumbar puncture (LP).

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
To describe the pharmacokinetics (PK) of AlpE in plasma and cerebrospinal fluid (CSF) in patients with newly diagnosed Tuberculosis Meningitis (TBM) | 15 days
  CSF/plasma ratio of alpibectir, ethionamide and the metabolite ethionamide sulfoxide

SECONDARY OUTCOMES:
To assess the safety and tolerability of alpibectir and ethionamide (Eto) in patients with TBM | 56 days
  Incidence of adverse events (AEs), including AEs ≥ grade 3, serious adverse events (SAEs), and AEs leading to AlpE discontinuation between D1 and D56

OTHER OUTCOMES:
To assess the effect of AlpE on the plasma PK of isoniazid (H), rifampicin (R), pyrazinamide (Z), ethambutol (E) (HRZE). | Day 15
  CSF/plasma ratio of HRZE
To assess the Mycobacterium tuberculosis (Mtb) culture conversion rate | 15 days
  To estimate the Mycobacterium tuberculosis (Mtb) culture conversion rate and time to detection (by MGIT), and cycle threshold (GeneXpert MTB/RIF Ultra) on the CSF and respiratory samples at screening, D3, and D15.